CLINICAL TRIAL: NCT03123146
Title: Functional Behavior-based Cognitive-Behavioral Therapy for Obsessive Compulsive Behavior in Children With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Cognitive Behavioural Therapy for Children With Autism Spectrum Disorder and Obsessive Compulsive Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tricia Vause (Other)
Collaborators: Ontario Mental Health Foundation (Other Government); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor-Investigator, Tricia Vause, Associate Professor, Brock University
Organization: Brock University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-066-VAUSE
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorder; Obsessive-Compulsive Behavior
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Autism Spectrum Disorder; Compulsive Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fb-Cognitive Behavioral Therapy (Experimental): Functional Behavior-Based Cognitive Behavioral Therapy: Group activities, individual work in parent-child dyads, group parent training, and social skills exercises.
  Interventions: Behavioral: Functional Behavior-Based Cognitive Behavioral Therapy
- Treatment as Usual (TAU) (No Intervention): Children assigned to this condition received "usual care," meaning that they could continue with any services. This group acted as a control group whereby access to intervention was patient-directed.

INTERVENTIONS:
Behavioral: Functional Behavior-Based Cognitive Behavioral Therapy — Fb-CBT involved nine 2-hour weekly sessions with three to four children in each group and two therapists. Therapy consisted of group activities, individual work in parent-child dyads, group parent training, and social skills exercises.
  Arms: Fb-Cognitive Behavioral Therapy

SUMMARY:
Individuals with high functioning autism spectrum disorder (ASD) frequently experience obsessions and/or compulsions that are similar to those specified in Diagnostic and Statistical Manual of Mental Disorders (5th ed.; DSM-5) criteria for obsessive compulsive disorder (OCD). However, little research exists on effective interventions for OCD symptoms (referred to as OCBs) in ASD. In a randomized controlled trial, a manualized functional behavior-based cognitive-behavior therapy (Fb-CBT) consisting of traditional CBT components (psychoeducation and mapping, cognitive-behavioral skills training, exposure, and response prevention) as well as function-based behavioral assessment will be evaluated. Participants will be assigned randomly to Fb-CBT or treatment as usual (TAU). Primary and secondary outcome measures will be used to evaluate the efficacy of the treatment, and will be administered at pre and post-intervention as well as six month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of ASD
* Presence of OCBs as defined by Sameness, Ritualistic and Compulsive subscales on the RBS-R
* a Full Scale IQ (WISC-IV; Wechsler, 2004) ≥ 70
* parent indicated no planned change in child medication during the study (unless the physician deemed the change medically necessary)

Exclusion Criteria:

* participation in treatment for anxiety
* participation in treatment for repetitive behaviour
* participation in treatment for intensive behavioural intervention

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Repetitive Behavior Scale (RBS_SCR) | Assessment occurred at baseline and 2 weeks following end of treatment, as well as at follow-up (6 months following the cessation of treatment)
  The RBS is a 43-item parent rating measure of repetitive behavior. It is comprised of a four-point Likert scale ranging from (0) behavior does not occur, to (3) behavior occurs and is a severe problem . The RBS_SCR scale specifically focusses on the assessment of sameness, compulsive, and ritualistic behaviors
Change in Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) | Assessment occurred at baseline and 2 weeks following end of treatment
  A 10-item, semi-structured interview used to assess symptom severity for children ages 6 through 17 years. Each item is rated on a 5-point ordinal scale from 0 (none) to 4 (extreme)' For the purpose of this study, only the 5-item Compulsion score was used pre and post-treatment.

SECONDARY OUTCOMES:
Change in Repetitive Behavior Scale 100 (RBS_100) | Assessment occurred at baseline and 2 weeks following the end of treatment, as well as at follow-up (6 months following the cessation of treatment)
  The final item on the RBS-R asks caregivers to rate on a scale from 1 to 100 how much OCBs affect the child and the people around them (1 is not a problem to 100 is as bad as can be imagined; Bodfish et al., 1999).
Change in The child Obsessive-Compulsive Impact Scale-Revised (COIS-R) | Assessment occurred at baseline and 2-weeks following the end of treatment, as well as at follow-up (6 months following the cessation of treatment)
  A 33-item, parent-report questionnaire that assesses OCD-related impairment in various areas of the child's life, including school, social, and home/family activities. For each item, the parent rates the child's level of impairment on a 4-point Likert scale from 0 (not at all) to 3 (very much).
Parent OCB Rating Scale. | Scale was completed by parents at baseline, each day throughout the 9-week treatment period, and at follow-up (6 months following the cessation of treatment)
  A Likert-type scale ranging from 1 (desired post-treatment levels of OCBs) to 3 (partial improvement from pre-treatment levels) to 5 (pre-treatment levels of OCBs) was used by parents to rate OCBs.

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Vause, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

REFERENCES:
- [Derived] Vause T, Jaksic H, Neil N, Frijters JC, Jackiewicz G, Feldman M. Functional Behavior-Based Cognitive-Behavioral Therapy for Obsessive Compulsive Behavior in Children with Autism Spectrum Disorder: A Randomized Controlled Trial. J Autism Dev Disord. 2020 Jul;50(7):2375-2388. doi: 10.1007/s10803-018-3772-x. PMID 30293128